CLINICAL TRIAL: NCT07249879
Title: A Phase 1, First-in-Human, Investigator-Initiated, Open-label Study to Assess the Safety, Feasibility, Cytokinetics, and Preliminary Antitumor Activity of GC511B in Adult Subjects With DLL3+ Relapsed/Refractory Small Cell Lung Cancer
Brief Title: This Study is an Open-lable, Phase I Study to Evaluate the Safety, Feasibility, Cytokinetics, and Preliminary Efficacy of GC511B in DLL3+ Relapsed/Refractory Small Cell Lung Cancer.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, NING LI, Ph.D. Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N6762000000
Record Dates: First submitted 2025-11-13; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Small Cell Lung Cancer
Keywords: Relapsed/Refractory Small Cell Lung Cancer;; DLL3+ expression; CAR-T cell therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages:
  Dose escalation stage: To determine MTD/MAD and evaluate the safety and tolerability of GC511B monotherapy.
  Dose expansion stage: To further determine RDE and evaluate the preliminary efficacy of GC511B monotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC511B CAR-T Cell Injection (Experimental): This study is a open-label clinical study. The main purpose is an IIT clinical trial to evaluate the safety and preliminary efficacy of GC511B dual CAR-T injection in Relapsed/Refractory Small Cell Lung Cancer subjects . The enrolled subjects were patients with DLL3+ Relapsed/Refractory Small Cell Lung Cancer (r/r SCLC) .
  Interventions: Drug: GC511B CAR-T Cell Injection

INTERVENTIONS:
Drug: GC511B CAR-T Cell Injection — This product is a lentiviral gene-modified autologous chimeric antigen receptor T-cell product that GC511B.Administration of GC511B CAR T-Cells a dose levels of DL1,DL2,DL3 and DL4 are administrated for each subject.Single IV infusion.

SUMMARY:
This is a First-in-Human, open-label, phase I dose-escalation clinical study to evaluate the safety and preliminary efficacy of GC511B CAR T cell injection in Adult with DLL3+ r/r SCLC subjects.

DETAILED DESCRIPTION:
This is a First-in-Human, open-label, phase I dose-escalation clinical study to evaluate the safety and preliminary efficacy of GC511B CAR T cell injection in Adult with DLL3+ r/r SCLC subjects.

this study consists of two parts: dose escalation and dose expansion: Dose Escalation: This part consists of two stages:Stage 1: Accelerated titration design to explore the effective starting dose;Stage 2: Bayesian optimal interval (BOIN) design to explore the MAD/MTD.The BOIN design will start with aDL1 as determined in Stage 1 and continue until either 9 subjects have been enrolled at a single dose level (DL) or the total number of subjects reaches 11.During the dose-escalation phase, following each dose level (DL) and/or scheduled dosing time point, the Safety Review Committee (SRC) will evaluate all adverse events (AEs), serious adverse events (SAEs), laboratory safety data from subjects in the DLT observation period, as well as all other relevant available data, to determine the next DL to be explored and/or dosing schedule and to provide recommendations for subsequent study conduct.

Dose expansion : The dose expansion phase will be initiated at the defined RDE to further investigate the safety, feasibility, CK, immunogenicity, PD, and preliminary antitumor activity of GC511B monotherapy and/or combination therapy. Up to 4 expansion cohorts may be opened to evaluate specific DLs and indications with up to 20 response-evaluable subjects included in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subject must be ≥ 18 years of age at the time of signing the ICF. Type of Subjects and Disease Characteristics
* 2.ECOG performance status 0-2.
* 3.Life expectancy ≥ 12 weeks.
* 4.At least 1 TL meeting RECIST v1.1 at baseline. Tumor assessment by CT scan or MRI must be performed within 28 days prior to apheresis.

  1. A lesion can be considered TL if the lesion previously subjected to radiotherapy has a clear boundary, is measurable as per RECIST v1.1, and has clear progression during or after the latest treatment;
  2. If a fresh biopsy sample is selected at screening from a tumor lesion, the tumor lesion should not be selected as a TL unless imaging is performed at least approximately 2 weeks after the biopsy to allow time for healing. In a case where there is only one measurable TL, caution should be taken when obtaining biopsy tissues during the treatment period.
* 5.Archival or representative tumor material for assessment of DLL3 expression levels can be provided.
* 6.Adequate organ function:

  a.Blood function: i.Hemoglobin ≥ 9 g/dL (without transfusion or erythropoietin therapy within 2 weeks prior to screening assessment); ii.Absolute neutrophil count ≥ 1.5×10^9/L and absolute lymphocyte count ≥ 0.6×10^9/L (without G-CSF use within 2 weeks prior to screening assessment);iii.Platelet count ≥ 75×10^9/L (without platelet transfusion or recombinant human thrombopoietin within 2 weeks prior to screening assessment).

  b.Hepatic function (based on normal values as defined by the clinical study site):i.Serum TBL ≤ 1.5 ×ULN;ii.ALT or AST ≤ 2.5×ULN in the absence of liver metastases; ALT and AST ≤ 5×ULN in the presence of liver metastases.

  c.Renal function (based on normal values as defined by the clinical study site): i.Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/minute calculated using the Cockcroft-Gault formula, or creatinine clearance ≥ 60 mL/minute calculated using 24-hour urine.ii.Urine protein <++. For subjects with proteinuria ≥ ++ on urine test paper at baseline, 24-hour urine must be collected and the content of protein in urine within 24 hours must be < 1 g.

  d.Coagulation function (based on normal values as defined by the clinical study site):i.PT≤1.5×ULN；ii.Thrombin time ≤ 1.5×ULN;iii.aPTT≤1.5×ULN。

  e.Cardiac function:i.New York Heart Association classification < class 3;ii.LVEF ≥ 50%.
* 7.Able to establish venous access and, in the judgment of the investigator, suitable for PBMC collection.
* 8.Women of childbearing potential must be non-lactating, and women of childbearing potential must have a negative result of highly sensitive serum pregnancy test during screening.
* 9.All subjects of childbearing age (including women of childbearing age and males with partners) must agree to take medically acceptable effective contraception measures as mentioned in Appendix G throughout the treatment period and for 2 years after the last CAR-T product reinfusion or until a negative CAR copy test, whichever occurs later.
* 10.Male subjects must agree not to donate sperm and female subjects must agree not to donate eggs throughout the treatment period and for 2 years after the last CAR-T product reinfusion or until a negative CAR copy test, whichever occurs later.
* 11.Capable of signing ICF (as mentioned in Appendix A), which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
* 12.The subject has provided ICF before starting any study-specific activity/procedure.
* 13.Able to communicate well with the investigator, and willing to comply with the study plan and able to complete the study as required.

Exclusion Criteria:

* 1.Pregnant or breastfeeding females, or female subjects with a positive pregnancy test result during the screening period (females not of childbearing potential are not required to receive a pregnancy test, such as metrectomy and/or bilateral oophorectomy, or amenorrhea for ≥ 12 months).
* 2.Subjects who have received a live vaccine within 4 weeks prior to initiation of apheresis or who plan to receive any vaccine (other than coronavirus disease 2019 vaccine) during the study.
* 3.Subject has a history of other acquired or congenital immunodeficiency; subject received organ transplant or bone marrow transplant.
* 4.The subject has a serious arterial/venous thromboembolic event or cerebrovascular accident within 6 months before apheresis, such as deep venous thrombosis (excluding asymptomatic and untreated muscle venous thrombosis), pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, and angina, except for lacunar infarction that is asymptomatic and does not require clinical intervention.
* 5.The subject has hereditary or acquired haemorrhage and thrombophilia (e.g., hemophilia, coagulation disorder, splenomegaly); the subject is receiving thrombolytic or anticoagulant therapy; the subject requires continuous antiplatelet therapy.
* 6.The subject has a QTc interval > 450 ms (males) or > 470 ms (females) during the screening period; the subject has a family or personal history of long or short QT syndrome; the subject has a history of clinically significant ventricular arrhythmias, or is currently receiving antiarrhythmic medication, or has a defibrillator implanted for arrhythmia.
* 7.The subject has other diseases that may seriously endanger the safety of the subject or affect the completion of the study, such as peptic ulcer, intestinal obstruction, intestinal paralysis, pulmonary fibrosis, renal failure, and uncontrolled diabetes.
* 8.The subject has an active or ongoing infection requiring systemic treatment (the subject may start study treatment 2 weeks after completion of anti-infective therapy).
* 9.History of any autoimmune nervous system disorder, including but not limited to: multiple sclerosis, neuromyelitis optica spectrum disorder, myasthenia gravis, Guillain Barre syndrome, and chronic inflammatory demyelinating polyradiculoneuropathy. Other active autoimmune or inflammatory disorders, including but not limited to inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), systemic lupus erythematosus, Sarcoidosis syndrome, granulomatosis with polyangiitis, autoimmune thyroid disease (Graves' disease) or rheumatoid arthritis. The following are exceptions to this criterion:

  1. The subject has vitiligo or autoimmune alopecia;
  2. The subject has autoimmune hypothyroidism (e.g., following Hashimoto's thyroiditis) and is stable on hormone replacement;
  3. Any chronic inflammatory or autoimmune skin disease that does not require systemic therapy;
  4. Subjects without active disease in the past 5 years may be enrolled in the study, but must first consult with the investigator;
  5. Subjects whose celiac disease is controlled by dietary management alone.
* 10.Subjects with known life-threatening hypersensitivity or other intolerance to cyclophosphamide or fludarabine, or severe allergic constitution; subjects with allergy to human serum albumin and dimethyl sulfoxide.
* 11.Active or chronic infectious diseases, including:

  1. HBV infection, defined as HBsAg positive or hepatitis B core antibody positive and HBV-DNA detectable;
  2. HCV infection, defined as HCV antibody positive and HCV-RNA detectable;
  3. HIV infection, defined as anti-HIV (1/2) positive;
  4. Syphilis infection, defined as TPPA positive with clinical or exposure evidence.
* 12.Prior receipt of anti-tumor therapies or participation in clinical studies;

  1. The subject has received prior CAR-T cell therapy or other gene-editing cell therapy;
  2. The subject participated in other clinical studies within 28 days prior to screening;
  3. Use of systemic corticosteroids (excluding inhaled corticosteroids) at a daily dose of ≥ 10 mg within 7 days prior to apheresis;
  4. Use of chemotherapy, radiotherapy, immunotherapy, or targeted therapy within 4 weeks or less than 5 drug half-lives, whichever is shorter, prior to apheresis;
  5. Subjects who have received traditional Chinese medicine treatment for a clear anti-tumor indication within 2 weeks before apheresis.
* 13.Toxicities from prior anticancer therapy that have not recovered to National Cancer Institute CTCAE v5.0 Grade 0 or Grade 1 (excluding alopecia, pigmentation, and other Grade ≤ 2 long-term toxicities considered irreversible by the investigator).
* 14.Subjects who previously discontinued administration due to adverse reactions such as immune-related pneumonitis, pituitary or thyroid dysfunction, or pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2026-11-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) Rate | 28 days
  DLT is defined as an AE that occurs within 28 days of GC511B CAR-T product reinfusion.DLT will be evaluated according to NCI-CTCAE V5.0 criteria
Adverse Events （AEs） | Up to 15 years from treatment discontinuation
  Proportion of subjects experiencing AE within 15 years after infusion of GC511B CAR-T cell injection.
Changes in vital signs to baseline | Up to 24 months from treatment discontinuation
  Include body temperature by CTCAE V5.0
Changes in Electrocardiogram(ECG) to baseline | Up to 24 months from treatment discontinuation
  ECG QT intervals
Changes in vital signs to baseline | Up to 24 months from treatment discontinuation
  Systolic and diastolic blood pressure by CTCAE V5.0
Changes in vital signs to baseline | Up to 24 months from treatment discontinuation
  Respiratory rate by CTCAE V5.0
Changes in vital signs to baseline | Up to 24 months from treatment discontinuation
  Pulse by CTCAE V5.0

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) | Up to 15 years from treatment discontinuation
  Cytokinetics (CK) profile of GC511B CAR-T celltherapy
Maximum plasma concentration (Cmax) | Up to 15 years from treatment discontinuation
  Cytokinetics (CK) profile of GC511B CAR-T celltherapy
Time to maximum plasma concentration (Tmax) | Up to 15 years from treatment discontinuation
  Cytokinetics (CK) profile of GC511B CAR-T celltherapy
Last detectable time point（Tlast） | Up to 15 years from treatment discontinuation
  Cytokinetics (CK) profile of GC511B CAR-T celltherapy
Last quantifiable concentratione (Clast) | Up to 15 years from treatment discontinuation
  Cytokinetics (CK) profile of GC511B CAR-T celltherapy
Replication-competent lentivirus(RCL) in peripheral blood | At baseline and within the selected time after the infusion of GC511B CAR-T cell
  RCL is monitored through mandatory viral testing
Objective Response Rate (ORR) | Up to 15 years study discontinuation
  ORR is defined as the percentage of subjects with confirmed CR or PR, and the denominator is defined as the number of subjects in the response evaluable set
Best Overall Response (BOR) | Up to 15 years study discontinuation
  BOR is defined as the best response a subject achieves based on evaluable data collected at all available time points prior to progression, or the last evaluable assessment result in the absence of disease progression or the initiation of subsequent anti-tumor therapy.
Duration of Response (DoR) | Up to 15 years study discontinuation
  DoR is defined as the time from the date of the first documented objective response (subsequently confirmed) to the first documented disease progression or death (for any reason in the absence of disease progression).
DCR at Week 8 | 12Weeks
  DCR at Week 8 is defined as the percentage of subjects who achieve and maintain a CR or PR at or prior to Week 8, or achieve SD and maintain for at least 4 weeks after CAR-T reinfusion.
Time to First Response（TTR） | Up to 15 years study discontinuation
  TTR is defined as the time from the date of CAR-T product reinfusion to the date of the first documented confirmed objective response that is subsequently confirmed
Percentage Change in Tumor Size | Up to 15 years study discontinuation
  Depth of tumor response is defined as the maximum percentage of shrinkage of TL compared with baseline.
Progression-free Survival(PFS) | Up to 15 years study discontinuation
  PFS is defined as the time from the date of CAR-T product reinfusion to the date of objective disease progression or death (all-cause death in the absence of progression).
Overall Survival(OS) | Up to 15 years study discontinuation
  OS is defined as the time from the date of CAR-T product reinfusion to the date of all-cause death, regardless of whether the subject receives another anti-tumor therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Gobroad Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No